CLINICAL TRIAL: NCT02238106
Title: A Single Dose, Placebo-controlled, Randomized, Double-blind, Double-dummy, Crossover Efficacy, Pharmacokinetics and Safety Comparison of Salmeterol Inhalation Powder (12.5 μg, 25 μg and 50 Salmeterol), Administered as the Xinafoate Salt From Hard Polyethylene Capsules Via the HandiHaler® 2, and Serevent® Diskus® (50 μg Salmeterol) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Salmeterol Inhalation Powder Administered as the Xinafoate Salt From Hard Polyethylene Capsules Via the HandiHaler® 2, and Serevent® Diskus® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.12
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

ARMS (5):
- Salmeterol inhalation powder, medium dose (Experimental): administered via HandiHaler®
  Interventions: Drug: Salmeterol medium dose; Drug: Placebo HandiHaler®; Drug: Placebo Diskus®
- Salmeterol inhalation powder, low dose (Active Comparator): administered via HandiHaler®
  Interventions: Drug: Salmeterol low dose; Drug: Placebo HandiHaler®; Drug: Placebo Diskus®
- Salmeterol inhalation powder, high dose (Active Comparator): administered via HandiHaler®
  Interventions: Drug: Salmeterol high dose; Drug: Placebo Diskus®
- Serevent® Diskus® (Active Comparator): administered via Diskus®
  Interventions: Drug: Serevent® Diskus®; Drug: Placebo HandiHaler®
- Placebo (Placebo Comparator): administered via Diskus® or HandiHaler®
  Interventions: Drug: Placebo HandiHaler®; Drug: Placebo Diskus®

INTERVENTIONS:
Drug: Salmeterol medium dose
  Arms: Salmeterol inhalation powder, medium dose
Drug: Salmeterol low dose
  Arms: Salmeterol inhalation powder, low dose
Drug: Salmeterol high dose
  Arms: Salmeterol inhalation powder, high dose
Drug: Serevent® Diskus®
  Arms: Serevent® Diskus®
Drug: Placebo HandiHaler®
  Arms: Placebo; Salmeterol inhalation powder, low dose; Salmeterol inhalation powder, medium dose; Serevent® Diskus®
Drug: Placebo Diskus®
  Arms: Placebo; Salmeterol inhalation powder, high dose; Salmeterol inhalation powder, low dose; Salmeterol inhalation powder, medium dose

SUMMARY:
The primary objective of this trial was to establish non-inferiority of lung function response to two doses [25 μg (1 capsule) and 50 μg (2 capsules of 25 μg)] salmeterol, administered as the xinafoate salt, in an inhalation powder delivered from hard polyethylene (PE) capsules via the HandiHaler® 2 compared to Serevent® Diskus® (salmeterol 50 μg, administered as the xinafoate salt) following single dose inhalation in patients with COPD. A hard capsule with half the strength (12.5 μg) was included to investigate a dose ordering effect.

The secondary objectives were to characterize the pharmacokinetics of salmeterol inhalation powder delivered by HandiHaler® 2 from the PE hard capsule(s) and salmeterol xinafoate delivered by Serevent® Diskus®, and to compare the safety of the different pharmaceutical forms and/or doses.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   * Patients must have relatively stable* airway obstruction with a pre-dose FEV1 ≤ 60% of predicted normal and FEV1 ≤ 70% of FVC at Visits 1 and 2

     * *The enrolment of patients who have had an exacerbation within six weeks prior to planned study entry should be postponed
3. At Visit 1, patients must demonstrate an improvement in FEV1 of ≥12% over the pre-bronchodilator value 45 minutes after inhalation of 4 puffs of 100 µg salbutamol (Sultanol® MDI)
4. Male or female patients 40 years of age or older
5. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years
6. Patients must be able to perform technically acceptable pulmonary function tests during the study period as required in the protocol
7. Patients must be able to inhale medication in a competent manner from the HandiHaler® 2 device and the Diskus® device

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with a recent history (i.e., six months or less) of myocardial infarction
3. Patients who have been hospitalized for heart failure (New York Heart Association (NYHA) class III or IV) within the past year
4. Patients with any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
5. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed
6. Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥600/mm3
7. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
8. Patients with known active tuberculosis
9. Patients with significant alcohol or drug abuse within the past two years
10. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1.
11. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program that will not be maintained throughout the duration of the study
12. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy
13. Patients who are being treated with antihistamines (H1 receptor antagonists), antileukotrienes or leukotriene receptor antagonists for asthma or excluded allergic conditions. See exclusion criterion No 6
14. Patients who have been treated with cromolyn sodium or nedocromil sodium within one month prior to Visit 1 or during the run-in period
15. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
16. Patients with known hypersensitivity to beta-adrenergics, lactose or any other components of the inhalation capsule delivery system or the Diskus®
17. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous three months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants, e.g.: Norplant®)
18. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Visit 1
19. Patients who have been treated with oral beta-adrenergics within one month prior to Visit 1 or during the run-in period
20. Patients who have been treated with theophylline preparations within one month prior to Visit 1 or during the run-in period
21. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®) within one month prior to Visit 1 or during the run-in period
22. Patients with any respiratory infections in the six weeks prior to the Screening Visit (Visit 1) or during the run-in period. In the case of a respiratory infection during the run-in period the latter may be extended up to six weeks
23. Patients who are currently participating in another study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change in area under the curve for the time period 0 to 12 hours (AUC0-12h) of the forced expiratory volume in one second (FEV1) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing

SECONDARY OUTCOMES:
Change in peak FEV1 | within 3 hours post-dosing
  Peak FEV1 is defined as the maximum FEV1 obtained within the first three hours post dosing
Change in peak forced vital capacity (FVC) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Change in FVC AUC0-12h | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Individual FEV1 measurements at each time point | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Individual FVC measurements at each time point | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Cmax (maximum measured concentration of the analyte in plasma) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
tmax (time from dosing to the maximum concentration of the analyte in plasma) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
λz (terminal rate constant in plasma) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
t½ (terminal half-life of the analyte in plasma) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
MRTih (mean residence time of the analyte in the body after inhalational administration) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | pre-dose and 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
Aet1-t2 (amount of analyte that is eliminated in urine from the time interval t1 to t2) | 0 to 3h 5min, from 3h 5min to 6h 5min, and from 6h 5min to 8h 5min after administration
fet1-t2 (fraction of administered drug excreted unchanged in urine from time point t1 to t2) | 0 to 3h 5min, from 3h 5min to 6h 5min, and from 6h 5min to 8h 5min after administration
CLR,t1-t2 (renal clearance of the analyte in plasma from the time point t1 to t2) | 0 to 3h 5min, from 3h 5min to 6h 5min, and from 6h 5min to 8h 5min after administration
Number of patients with adverse events | up to 36 days

REFERENCES:
- See also: Related Info — http://clintriage.rdg@boehringer-ingelheim.com